CLINICAL TRIAL: NCT02292316
Title: Falls With Fracture : Role of Cognitive Disorders and Comparison With Bone Fragility
Acronym: CFC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RCB 2011A00556-35
Record Dates: First submitted 2014-09-26; First posted 2014-11-17 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Accidental Falls; Fractures
Keywords: middle-aged and aged adults; fall in the previous year
MeSH Terms: conditions — Fractures, Bone | interventions — Gait; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fall with fracture (Experimental): Fall with fracture in the last 6 months; Interventions : behavioral, biological and other; Behavioral intervention includes gait and cognitive assessments Blood sample Osteodensitometry
  Interventions: Behavioral: gait and cognitive assessments; Biological: blood sample; Other: osteodensitometry
- controls (Sham Comparator): Fall without fracture in the last 12 months; Interventions : behavioral, biological and other; Behavioral intervention includes gait and cognitive assessments Blood sample Osteodensitometry
  Interventions: Behavioral: gait and cognitive assessments; Biological: blood sample; Other: osteodensitometry

INTERVENTIONS:
Behavioral: gait and cognitive assessments — several tests are given in each domain
Biological: blood sample — routine analyses in rheumatology such blood count and 25OH-D
Other: osteodensitometry — Looking for osteoporosis

SUMMARY:
The purpose of this study is to determine whether cognitive disorders are a risk factor for a fracture after a fall independently of a bone fragility.

DETAILED DESCRIPTION:
The fall is a major problem in the elderly. After 65 year old, falls represent 84% of daily living accidents and almost half of the post fall injuries are fractures (Ricard and Thélot, 2007). These falls with fracture lead to a loss of autonomy and a high health cost. Their prevention is a crucial focus of research.

Even if it is obvious that subjects with osteoporosis have a higher risk of fracture than those with a normal bone mineral density, recent studies have shown that most victims of fracture post-fall do not comply with the densitometric definition of osteoporosis.

It is well established that the presence of cognitive disorders, frequent in the elderly, is an important risk factor for falls; It might also be a risk factor for fracture after a fall with an unadapted postural or balance control.

The investigators will test this hypothesis on 150 victims of fracture (upper or lower limb) consecutive to a fall from standing height, recruited in the hospitals of Caen and Rouen (France) in the context of their medical follow-up (with blood and dual energy x-ray absorptiometry [DXA] exams). These patients will be matched to 150 control participants (victims of a fall with no fracture, submitted to the same exams).

All the participants are subjects to an in-depth study of cognitive functions, postural and walking tests and to various scales (daily life activities, depression, ...).

These exams will take half a day, with a two-year follow up (in which the participant will have to note new falls and new medical treatments)

ELIGIBILITY:
Inclusion Criteria:

* Affiliation to the social security system
* For subjects with fracture : victim of a low-energy fracture of the upper or lower limb that was consecutive to a fall from standing height, and who has accepted to realize a DXA exam in the context of the medical follow-up
* For control subjects : victim of a fall from standing height, with no fracture, matched in terms of age, sex, socio-cultural level and living space with subjects with fracture.
* Written informed consent

Exclusion Criteria:

* Subject who is deprived of liberty, under supervision or legal guardianship
* Pathology affecting balance (Parkinson's disease, after-effects of stroke, …)
* Important visual impairment : age-related macular degeneration, …
* Depressed state
* Important consumption of alcohol (> 14 drinks per week for women / >21 for men)
* Subject who is concurrently participating in another clinical study (unless prior notice of the principal investigator)
* Fall has been caused by a third party (e.g. : pushing), is not from standing height (e.g. : fall from a ladder); fracture is not a low-energy one (e.g. : further a fall during running)
* For subjects with fracture :

  * The fracture is not consecutive to a fall
  * The fracture is pathological, beyond osteoporosis (e.g. : bone metastases)
  * The last fall responsible for a fracture goes back more than 6 months
* For control subjects :

  o The fall goes back more than 12 months
* The fall has led to a medical consultation

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2011-11-15 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Analysis of a global cognitive efficiency score Analysis of bone mineral density | on the inclusion day and two years after
  MMS, MoCA

SECONDARY OUTCOMES:
Age | on the inclusion day and over two years
Cognitive scores | on the inclusion day and over two years
  Mainly tests of memory, attention and executive functions
Fracture features | on the inclusion day and over two years
  Location and severity
Balance and walking parameters | on the inclusion day and over two years
  Tinetti scale, TUG and dual-tasks
handgrip force | on the inclusion day and over two years
  using a dynamometer
Daily life scales scores | on the inclusion day and over two years
  Mainly IADL
fear of falling | on the inclusion day and over two years
  ABC-scale
functional restrictions score | on the inclusion day and over two years
  Lequesne score
Degree of depression | on the inclusion day and over two years
  MADRS
biological data | on the inclusion day and over two years
  25OHD
Dual-energy X-ray absorptiometry | on the inclusion day and two years after
  bone mineral densitometry

CONTACTS AND LOCATIONS:
Overall Officials: Christian Marcelli, Professor, Principal Investigator — CHU of Caen
Locations (2):
- France (2):
  - University Hospital, Caen
  - Dr Alain Daragon, Rouen

REFERENCES:
- [Derived] Langeard A, Pothier K, Chastan N, Marcelli C, Chavoix C, Bessot N. Reduced gait and postural stability under challenging conditions in fallers with upper limb fracture. Aging Clin Exp Res. 2019 Apr;31(4):483-489. doi: 10.1007/s40520-018-0992-z. Epub 2018 Jul 4. PMID 29974390
- [Derived] Langeard A, Pothier K, Morello R, Lelong-Boulouard V, Lescure P, Bocca ML, Marcelli C, Descatoire P, Chavoix C. Polypharmacy Cut-Off for Gait and Cognitive Impairments. Front Pharmacol. 2016 Aug 31;7:296. doi: 10.3389/fphar.2016.00296. eCollection 2016. PMID 27630572